CLINICAL TRIAL: NCT05749211
Title: Efficacy and Safety of Huaier Granule in Combination With Nilaparil in First-line Maintenance Therapy in Postoperative Patients With Stage III/IV BRCA Wild-type Ovarian Cancer: a Single-center Prospective, Single-arm Study
Brief Title: Huaier Granule in Combination With Nilaparil in Therapy Patients With Stage III/IV BRCA Wild-type Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023(02)
Record Dates: First submitted 2023-01-19; First posted 2023-03-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Huaier granule (Experimental): Huaier granule is supplied as 20-g granule. Huaier granule will be administered as 20 g orally tid x 28 days (continuous). One cycle = 28 days. There is no planned treatment interruption between cycles. In the absence of intolerable toxicity, a patient may continue to receive treatment with Huaier granule until disease progression, or until 24 months have elapsed.
  Interventions: Drug: Huaier granule

INTERVENTIONS:
Drug: Huaier granule — Oral administration, 20 g once, 3 times a day, continued until progression or intolerance of toxicity
  Other Names: Niraparib

SUMMARY:
This is a single-center, prospective, single-arm clinical trial to evaluate the efficacy and safety of Huaier granules in combination with immunotargeted agents in postoperative patients with ovarian cancer.

DETAILED DESCRIPTION:
Primary objective :

1) To evaluate the efficacy of Huaier granule combined with immunotargeted drugs in the treatment of postoperative ovarian cancer patients

Secondary objectives:

1)To analyze the safety of Huaier granule in the treatment of postoperative ovarian cancer patients; 2)2) To analyze the influence of Huaier granule on postoperative quality of life of patients with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* According to FIGO criteria, participants must have a histological diagnosis of high-grade serous or endometrioid carcinoma, or high-grade serous or endometrioid predominantly ovarian, fallopian tube cancer, or stage III or IV primary peritoneal carcinoma
* Inoperable stage III and IV patients; All stage III and IV patients who can accept initial or intermittent tumor reduction surgery, regardless of the residual lesion status after surgery
* Patients who had undergone abdominal chemotherapy; All participants must undergo 6 and 9 cycles of platinum-based therapy; Participants were required to receive 2 cycles of postoperative platinum therapy following interphase tumor reduction surgery; Participants had to be assessed by a physician for complete response (CR) or partial response (PR) after 3 cycles of treatment; Participants had to have cancer antigen 125 (CA-125) within the normal range or ca-125 decreased by more than 90%(%) to be stable during their first-line therapy
* All participants must agree to be tested for central tumor BRCA
* Fertile participants must have a negative serum or urine pregnancy test (human chorionic gonadotropin [hCG]) within 7 days of receiving the first dose of study treatment.

Exclusion Criteria:

* Participants had epithelial ovarian carcinosarcoma or mucinous or clear cell subtypes of undifferentiated ovarian cancer
* The participants had already undergone more than two tumor-reduction surgeries for the study disease
* Participants became pregnant or lactated or expected to become pregnant during study treatment and 180 days after the last dose of study treatment
* Participants were known to be allergic to the ingredients or excipients of the study drug
* Participants had previously been treated with a known PARP inhibitor or had participated in any treatment group that included the use of a known PARP inhibitor
* Participants received bevacizumab maintenance therapy
* Subjects received investigational therapy within 4 weeks or at intervals not exceeding 5 investigational drug half-lives, whichever is longer, prior to the study's first scheduled dosing date
* Participants had known grade 3 anemia, neutropenia or thrombocytopenia that persisted due to prior chemotherapy. 4 weeks；
* Throughout the study treatment period, participants were treated with conditions (such as transfusion-dependent anemia or thrombocytopenia) or laboratory abnormalities that could confound study results or interfere with their participation, including:

  * Participants received blood transfusions (platelets or red blood cells) within 2 weeks of the first dose of study treatment
  * Participants received colony stimulating factor (e.g., granulocyte-colony-stimulating factor [G-CSF] or recombinant erythropoietin) within 2 weeks prior to the first dose of study treatment;
* Participants had been diagnosed and/or treated for invasive cancer less than 5 years prior to enrollment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival (PFS) | up to 2 years from start of treatment
  PFS according to the RECIST 1.1 criteria, based on the investigator's assessment.

SECONDARY OUTCOMES:
Median Progression Free survival | Every 3 month until 2 years from start of treatment
  mPFS is defined as the median time from study entry to date of first documented objective tumor recurrence according to RECIST 1.1
1-year progression-free survival rate | up to 1 years
  The time from study entry to the time of disease progression as determined by the investigator (by clinical, radiological or pathological means) or death from any cause
Median overall survival | Every 3 month until 2 years from start of treatment
  Median observed length of life from entry into the study to death; or for living patients, the date of last contact regardless of whether or not this contact is on a subsequent protocol
1 year overall survival rate | 1 year
  Observed length of life from entry into the study to death; or for living patients, the date of last contact regardless of whether or not this contact is on a subsequent protocol.
overall survival | From study entry to death or last contact, up to 2 years of follow-up
  OS is defined as the time from start of treatment to date of death due to any cause, or last patient contact
Quality of life score（ EQ-5D） | Every 3 month until 2 years from start of treatment
  questionnaires to be completed by patients and collected frequently during the trial
Quality of life score（EORTC-QLQ-OV28） | Every 3 month until 2 years from start of treatment
  Assessment of quality of life according to the QLQ-OV28/EORTC scales
Quality of life score（EORTC-QLQ-C30） | Every 3 month until 2 years from start of treatment
  Assessment of quality of life according to the QLQ-C30/EORTC scales
Quality of life score（FACT-O） | Every 3 month until 2 years from start of treatment
  The FACT-O questionnaire consists of a Physical Well-Being Section, Social/Family Well-Being Section, Emotional Well-Being Section, Functional Well-Being Section, and Additional Concerns Section
the rates of AEs and SAEs | up to 2 years
  frequency of adverse events according to MedDRA terms